CLINICAL TRIAL: NCT04435964
Title: Gender Difference in sidE eFfects of ImmuNotherapy: a Possible Clue to Optimize cancEr tReatment
Acronym: G-DEFINER
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Karolinska University Hospital (Other); St Vincent's University Hospital, Ireland (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: INT156-19
Record Dates: First submitted 2020-06-11; First posted 2020-06-17 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2021-09

CONDITIONS: Melanoma; Lung Cancer; Head and Neck Cancer; Urogenital Neoplasms; Breast Cancer
MeSH Terms: conditions — Melanoma; Lung Neoplasms; Head and Neck Neoplasms; Urogenital Neoplasms; Breast Neoplasms | interventions — Immunotherapy; Drug Therapy; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Gene-expression analysis. Blood samples will be taken in order to identify immune-related genes in patients with various solid tumors treated with ICI associated with the development of irAEs.
  * SNPs analysis. Blood samples will be taken in order to perform a preliminary genome wide association study for the identification of germline variations associated with the development of irAEs. with the hypothesis that the individual's genetic makeup may be related to irAEs.
  * Microbiome analysis. Stool collection will be performed to analyze gut microbiota aiming at performing RNA/DNA sequencing analysis for identifying components associated with the development of irAEs.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overall series: Patients treated with immunocheckpoint inhibitors (ICI) irrespective of treatment schedule. No limitations to previous lines of treatment. ICI therapy may be either as single agent or in combination. Concomitant chemotherapy (CT) and radiotherapy (RT) is allowed.
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Drug: Immunotherapy — Patients treated as per clinical prescription with immunocheckpoint inhibitors (ICI) irrespective of treatment schedule, either as single agent or in combination with chemotherapy and/or radiotherapy
  Other Names: Chemotherapy; Radiotherapy

SUMMARY:
The study aim is to investigate the differences between sex and gender in the immune-related adverse events (irAEs) development associated with immune checkpoint inhibitors (ICI) treatment. The study will be a multicenter prospective observational study focusing on biological differences between females and males, possibly affecting discrepant irAEs incidence.

DETAILED DESCRIPTION:
The study aim is to investigate the differences between sex and gender in the immune-related adverse events (irAEs) development associated with immune checkpoint inhibitors (ICI) treatment.

In common feeling, sex and gender represent the same concept, that is the traditional division of individuals into females (F) and males (M) defined by differential organization of chromosomes, reproductive organs, and sex steroid levels. However, if going beyond these aspects, which characterize "sex", it can be observed how the differences between people are also characterized by behaviors and relationships that are the product of the culture and sociality typical of human beings. This is what is called "gender", i.e. the process of social and cultural construction that determines the behaviors that give life to the status of an individual. Gender is therefore learned and not innate. Sex and gender do not constitute two opposing but interdependent dimensions: the process of determining gender identity is triggered on biological characters. The relationship between sex and gender varies according to geographical areas, historical periods and cultures.

Sex influences the adaptive immunity, and may influence irAEs types, frequency and severity. Together with genetic and biological differences, the roots of irAEs inequalities between F and M could be linked to psycho-social and behavioral determinants. IrAEs usually develop within the first few weeks to 6 months after treatment initiation; however, they can also present after cessation of ICI therapy. Most studies indicate that prolonged treatment does not result in an increased cumulative incidence of irAEs. Accumulating evidences support the existence of sex-driven differences in immune responses as potential factors contributing to disease outcome and response to therapy. Increasing use of ICI is associated with immune-related adverse events caused by non-specific activation of the immune system.

The investigators will conduct a multicenter prospective observational study investigating sex differences in irAEs in relation to clinical factors and genetic, immunological and hormonal profiles. By focusing on biological F/M differences possibly affecting discrepant irAEs incidence, sex inequality will be explicitly addressed and complemented by the exploration of association between gender dimension and irAEs development. Exploring the irAEs occurrence in a "real world" (outside RCT) context will be more easily translated in a ready-to-use personalized approach to irAEs timely diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Histologically confirmed diagnosis of one of the following cancers: melanoma, lung, head and neck, urogenital, breast cancer. In addition, other solid tumors characterized by the presence of microsatellite instability (MSI-high), treated with immunocheckpoint inhibitors (ICI) irrespective of treatment schedule. It is possible to include patients treated with Immunotherapy in a compassionate use setting.
* Any disease stage.
* Patients eligible for immune checkpoint inhibitors (ICI)-containing regimens: ICI single agent; Combination of ICIs; ICI-chemotherapy combination; ICI-radiotherapy combination.
* Any treatment setting (neoadjuvant, adjuvant, advanced disease, maintenance).
* Patient age ≥18 years
* ECOG Performance Status of 0-2.
* Adequate bone marrow, liver and renal function.
* Life expectancy of at least 12 weeks.

Exclusion Criteria:

* Patients not eligible for ICI-containing regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To allow for balanced sex groups, we will include patients according to the following stratification : ICI: 100 F/100 M; ICI+ CT/RT: 100 F/100 M. Due to the current ICI use in clinical practice we are expecting to mainly populate the ICI strata during the first recruitment period. As the recruitment progresses, the sample will be enriched of ICI+CT and ICI+RT treated patients, since combinations are expanding for many cancers such for instance melanoma, lung and head and neck
Sampling Method: Non-Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Immune-related severe (G≥ 2) adverse events (irAEs) | 1 year
  The incidence of first severe (G≥ 2) irAEs of any type will be estimated in females and males

SECONDARY OUTCOMES:
Immune-related adverse events (irAEs) | 1 year
  The incidence of irAEs of any type and any grade will be estimated in females and males

CONTACTS AND LOCATIONS:
Overall Officials: Rosalba Miceli, PhD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT04435964/Prot_SAP_000.pdf